CLINICAL TRIAL: NCT03241654
Title: Decreasing Trigger Sensitivity Could Assist PEEP to Further Improve Regional Aeration and Homogeneity During Pressure Assist Ventilation: A Preliminarily Physiological Study
Brief Title: Decreasing Trigger Sensitivity Could Assist PEEP to Further Improve Regional Ventilation Distribution
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY-2017-001
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-08

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the lowest trigger sensitivity: The flow trigger of ventilator was set as the lowest level of sensitivity.
  Interventions: Procedure: flow trigger
- the highest trigger sensitivity: The flow trigger of ventilator was set as the highest level of sensitivity.
  Interventions: Procedure: flow trigger

INTERVENTIONS:
Procedure: flow trigger — The flow trigger will be adjust during the pressure assist ventilation.

SUMMARY:
In mechanically ventilated patients during supine position, alveolar collapse usually distributes in dependent lung region.Decrease of flow trigger sensitivity might improve homogeneous of tidal volume distribution.

DETAILED DESCRIPTION:
In mechanically ventilated patients during supine position, alveolar collapse usually distributes in dependent lung region. High positive end expiratory pressure (PEEP) has been applied to improve the homogeneous distribution of ventilation by increasing the end expiratory lung ventilation (EELV) and alveolar recruitment. However, for patients who increasing PEEP in some extent still existed poor aeration in the dependent region, further elevating PEEP seems to be unreasonable that perhaps lead to overdistension. Decreasing trigger sensitivity might further evoke inspiratory efforts to improve the ventilation for this type of patients.The Electrical impedance tomography (EIT) was applied in monitoring the regional ventilation distribution at the bedside.

ELIGIBILITY:
Inclusion Criteria:

1. The post operative patients who received pressure support ventilation;
2. After the clinical PEEP was evaluated 5cmH2O, the tidal volume distribution still existed heterogeneity.

Exclusion Criteria:

1. Under 18 years;
2. History of diaphragm dysfunction and surgery;
3. Central respiratory drive dysfunction;
4. history of esophageal, gastric or lung surgery;
5. The contraindication of using EIT (pacemaker, defibrillator, and implantable pumps).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The postoperative patients receiving pressure support ventilation and existing heterogenous ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
The homogeneity of distribution of tidal volume | within 20 minutes after changing flow trigger
  EIT was used to monitoring the homogeneity of distribution of tidal volume that was divided into two contiguous regions of interest (ROI) equally, the dependent and non-dependent area. The ratio of relative distribution of tidal ventilation of two ROI was calculated.

SECONDARY OUTCOMES:
Changes in global and regional EELV | within 20 minutes after changing flow trigger
  The change of EELV was measured after changing flow trigger based on the baseline level.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Jian-Xin Zhou, Beijing, Beijing Municipality, China